CLINICAL TRIAL: NCT07167433
Title: Ovarian Cancer Epidemiology and Care in Brazil: A Multicenter Perspective (OLIVIA Study) Observational, Bi-directional (Prospective and Retrospective) Study for Patients With Newly Diagnosed Ovarian Cancer Stages IA to IVB, or Persistent or Recurrent Disease From January 2021; Irrespective of Histology
Brief Title: Observational, Bi-directional (Prospective and Retrospective) Study for Patients With Newly Diagnosed Ovarian Cancer Stages IA to IVB, or Persistent or Recurrent Disease From January 2021; Irrespective of Histology
Acronym: OLIVIA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00051
Record Dates: First submitted 2025-08-18; First posted 2025-09-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: patients newly diagnosed with ovarian cancer across stages IA to IVB, and those with persistent or recurrent disease, diagnosed from January 2021 onwards

SUMMARY:
The findings from this study have the potential to serve as a foundation for evaluating the current practices related to surgical procedures, systemic therapies, hyperthermic intraperitoneal chemotherapy, and referrals to geneticists for OC patients. By identifying the strengths and weaknesses of the existing care, this project intends to generate valuable insights that can lead to the implementation of quality parameters for the treatment of ovarian cancer in the country.

DETAILED DESCRIPTION:
This study is an observational, bi-directional (prospective and retrospective) analytical study designed to assess the sociodemographic, clinical, and pathological characteristics of patients with ovarian cancer, stages IA to IVB, as well as those with persistent or recurrent disease. The study will include 250 patients who meet the eligibility criteria of being 18 years or older, with a diagnosis of ovarian cancer from January 2021, irrespective of histology, over a 1-year enrollment period across 20 participating sites.

Upon enrollment, baseline data will be collected, which includes sociodemographic details, clinical information, pathological findings, and genetic testing and counseling data. Follow-up data will be gathered at 12, 24, and 36 months to monitor treatment patterns and outcomes. These data collection points will allow for the evaluation of both short-term and long-term outcomes, providing valuable insights into the progression and management of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old;
* Newly diagnosed ovarian cancer stages IA to IVB, or persistent or recurrent disease from January 2021;
* Irrespective of histology

Exclusion Criteria:

* Borderline tumors;
* Pregnancy;
* Synchronous tumor or second primary in the last 5 years (except thyroid cancer and non-melanoma skin cancer);

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study base consists of patients newly diagnosed with ovarian cancer across stages IA to IVB, and those with persistent or recurrent disease, diagnosed from January 2021 onwards. The study will span 20 research sites across diverse geographical locations, ensuring a broad representation of different healthcare settings and patient demographics. The study population will include patients aged 18 years and older, irrespective of histological subtype. Over a 12-month enrollment period, a total of 250 patients are expected to be included in the study. The follow-up period will extend for 3 years, with data collection occurring at 12, 24, and 36 months.
Study Population: The study base consists of patients newly diagnosed with ovarian cancer across stages IA to IVB, and those with persistent or recurrent disease, diagnosed from January 2021 onwards.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Description of socio-demographic characteristics | Throught study a completation, an average of 3 years
  The study's findings could provide a basis for evaluating current practices in ovarian treatment and other characteristics about this disease.
  By identifying strengths and weaknesses in existing care, the project aims to offer insights that may lead to the implementation of quality parameters for ovarian cancer treatment in the country.
  No formal statistical comparisons are begin performed for the primary outcomes of this study.
Description of pathological characteristics | Throught study a completation, an average of 3 years
  The study's findings could provide a basis for evaluating current practices in ovarian treatment and other characteristics about this disease.
  By identifying strengths and weaknesses in existing care, the project aims to offer insights that may lead to the implementation of quality parameters for ovarian cancer treatment in the country.
  No formal statistical comparisons are being performed for the primary outcomes of this study.
Description of treatment | Throught study a completation, an average of 3 years
  The study's findings could provide a basis for evaluating current practices in ovarian treatment and other characteristics about this disease.
  By identifying strengths and weaknesses in existing care, the project aims to offer insights that may lead to the implementation of quality parameters for ovarian cancer treatment in the country.
  No formal statistical comparisons are being performed for the primary outcomes of this study.

SECONDARY OUTCOMES:
Treatment interval of systemic therapy in metastatic disease | Throught study a completation, an average of 3 years
  The study's findings could provide a basis for evaluating current practices in ovarian treatment and other characteristics about this disease.
  By identifying strengths and weaknesses in existing care, the project aims to offer insights that may lead to the implementation of quality parameters for ovarian cancer treatment in the country.
  No formal statistical comparisons are beign performed for the outcomes of this study.
Disease free-survival | Throught study a completation, an average of 3 years
  The study's findings could provide a basis for evaluating current practices in ovarian treatment and other characteristics about this disease.
  By identifying strengths and weaknesses in existing care, the project aims to offer insights that may lead to the implementation of quality parameters for ovarian cancer treatment in the country.
  No formal statistical comparisons are beign performed for the outcomes of this study.
Time to next chemotherapy | Throught study a completation, an average of 3 years
  The study's findings could provide a basis for evaluating current practices in ovarian treatment and other characteristics about this disease.
  By identifying strengths and weaknesses in existing care, the project aims to offer insights that may lead to the implementation of quality parameters for ovarian cancer treatment in the country.
  No formal statistical comparisons are beign performed for the outcomes of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/